CLINICAL TRIAL: NCT01546324
Title: Prenatal Diagnosis of Fetal DNA Isolated From Maternal Plasma
Brief Title: Collection of Maternal Blood Samples for Development of Non-invasive Prenatal Diagnostic Testing
Status: Completed | Type: Observational
Sponsor: Natera, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IVF013
Record Dates: First submitted 2012-02-24; First posted 2012-03-07 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2013-08

CONDITIONS: Pregnancy Following IVF With PGS/PGD
Keywords: Maternal Blood; PGD; PGS; Natera; Gene Security Network; Non-invasive prenatal diagnosis
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant women: Women pregnant following the use of Natera's PGS/PGD testing
  Interventions: Procedure: Blood draw

INTERVENTIONS:
Procedure: Blood draw — Maternal blood draw at approximately 8-17 weeks gestation.

SUMMARY:
The purpose of this study is to collect blood samples from pregnant women who achieved pregnancy following in-vitro fertilization (IVF) with Natera's preimplantation aneuploidy screening (with or without single gene gene testing). These samples will be used for test development of non-invasive prenatal diagnostic testing.

DETAILED DESCRIPTION:
Eligible subjects will sign a consent form and have blood drawn at approximately 8-17 weeks gestation. Subjects will received $200 reimbursement for providing this blood sample. The collected samples will be used to help develop non-invasive prenatal diagnostic testing using Natera's Parental Support technology which is already commercialized for genetic diagnosis of in-vitro embryos. In this study, the technology will be tested for it's ability to analyze fetal-specific pieces of DNA isolated from the mother's blood. No results of the maternal blood testing will be reported to the subject or to their physicians.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women willing to donate a blood sample during the first or second trimester of their pregnancy (approximately 8-17 weeks gestation)
* Use of Natera (formerly Gene Security Network)'s commercial preimplantation genetic testing (PGS/PGD)to achieve the current pregnancy

Exclusion Criteria:

* Pregnant women who did not use Natera (formerly Gene Security Network)'s PGS/PGD testing to achieve their current pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women 18 years of age or older who used Natera (formerly Gene Security Network)'s Preimplantation Genetic testing (PGS/PGD) to achieve their current pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2012-02; Primary Completion 2012-05 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Collection of 500 maternal blood samples to be used for development of non-invasive prenatal diagnostic testing. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Rabinowitz, PhD, Principal Investigator — CEO, Natera, Inc
Locations (1):
- Natera, Inc, Redwood City, California, United States